CLINICAL TRIAL: NCT02849223
Title: Transcranial Direct Current Stimulation (TDCS) as an Intervention for Patients With Traumatic Brain Injury
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: State of Minnesota (Unknown); Minnesota Veterans Medical Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Tasha Nienow, Staff Psychologist, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4654-A
Record Dates: First submitted 2016-07-24; First posted 2016-07-29 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-06

CONDITIONS: Traumatic Brain Injury
Keywords: Mild Traumatic Brain Injury; Transcranial Direct Current Stimulation; Working Memory
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Direct Current Stimulation (Experimental): Participants will receive 24 sessions (2 times a week) of anodal transcranial direct current stimulation concurrent with working memory training. Stimulation will be administered at 2 milliamps (mA) for 20 minutes over the left dorsal lateral prefrontal cortex.
  Interventions: Device: Anodal Transcranial Direct Current Stimulation
- Sham (Sham Comparator): Participants will receive 24 sessions of working memory training. The experience of transcranial direct current stimulation will be simulated by administering 30 seconds of stimulation at the beginning of the session.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Anodal Transcranial Direct Current Stimulation — 2 milliamps (mA) of anodal stimulation will be applied to the left dorsal lateral cortex for 20 minutes concurrent with working memory training.
  Arms: Transcranial Direct Current Stimulation
Device: Sham stimulation — 30 seconds of anodal TDCS stimulation will be applied to the left dorsal lateral cortex concurrent with working memory training
  Arms: Sham

SUMMARY:
The primary aim of this study is to assess the magnitude of transcranial direct current stimulation (tDCS) -induced cognitive and functional change in patients with mild traumatic brain injury. This study will also attempt to identify biomarkers associated with treatment response. Last, acceptability and tolerability of procedures will be assessed. To accomplish these aims, a randomized, double-blind, sham-controlled, parallel groups, pilot study will be conducted in which participants are assigned to 24 sessions of tDCS or sham stimulation offered concurrent with working memory training. Neural efficiency will be measured with electroencephalogram (EEG) pre and post-intervention.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a safe, non-invasive neuromodulation technique that shows promise as an intervention technique. The primary aim of this study is to assess the magnitude of tDCS-induced cognitive and functional change in patients with mild traumatic brain injury (TBI). In this double-blind, sham-controlled, pilot study, 24 veterans with mild TBI will be randomized to tDCS or sham conditions. Stimulation will be administered with a StarStim neurostimulator at 2 milliamps (mA) for 20 minutes. The anodal electrode will be placed over the left dorsal lateral prefrontal cortex. Twenty-four sessions of stimulation will be administered concurrent with 20 minutes of working memory training. Participants will continue with an additional 40 minutes of working memory training post-stimulation. Participant experience with neuromodulation will be assessed with a self-report questionnaire that lists common reactions to tDCS. Participant perception of the value of neuromodulation procedures will be assessed at weeks 4 and 8. A second aim is to identify biomarkers of treatment response. Resting state electroencephalogram (EEG) will be collected at three time points: prior to the first tDCS training session, immediately after the first training session, and post-intervention. This study will provide preliminary evidence of the efficacy of providing tDCS as an intervention to enhance cognitive and functional outcomes for individuals with mild traumatic brain injury. Furthermore, the results of this study will also increase the understanding of the mechanisms by which tDCS enhances cognitive performance. This knowledge has the potential to provide insight into the underlying therapeutic process as well as to guide development of the next generation of interventions. In addition, acceptability of the intervention will be monitored to identify potential barriers to administering tDCS in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled at the Minneapolis Veterans Affairs (VA) Health Care System
* Age of 18 and 65
* Sustained a mild traumatic brain injury more than 1 year ago.

Exclusion Criteria:

* Presence of a psychotic disorder
* Severely depressed
* Clinically unstable due to a hospitalization or medication change in the previous 4 weeks
* Mild substance use disorder in the last month
* Moderate to Severe substance use disorder in the last six months
* Behavioral problems that prevent participation in a group intervention
* Premorbid intellectual ability (IQ) below 70
* Unable to provide informed consent
* Have a guardian of person
* Have another existing neurological condition that impacts cognitive functioning
* Not fluent enough in English to understand testing procedures
* Have a medical condition that is incompatible with transcranial direct current stimulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Wechsler Adult Intelligence Scale (WAIS)-III Working Memory Index | Post-Intervention, 12 weeks after baseline assessment
  Standard score

SECONDARY OUTCOMES:
University of California Performance Based Skills Assessment | Post-Intervention, 12 weeks after baseline assessment
  Total Score

CONTACTS AND LOCATIONS:
Overall Officials: Tasha M Nienow, PhD, Principal Investigator — Minneapolis Veteran Affairs Health Care System
Locations (1):
- Minneapolis Veterans Affairs Health Care System, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No